CLINICAL TRIAL: NCT02491021
Title: Outpatient Based Physical Rehabilitation for Survivors of Prolonged Critical Illness - a Randomised Controlled Trial
Brief Title: Outpatient Based Physical Rehabilitation for Survivors of Prolonged Critical Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David McWilliams, Mr David McWilliams, University Hospital Birmingham NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Q1402/39
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Rehabilitation After Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): Treatment Group (TG) The TG underwent a 7-week outpatient rehabilitation programme comprising both exercise and education sessions under the direct supervision of the physiotherapy team. The exercise intervention was 20 minutes, 3x/week (1 supervised, 2 self directed) titrated to a specific intensity based on risk stratification - highvs low risk). The intervention also included 6 x 1 hour education sessions.
  Interventions: Other: Rehabilitation Class
- Control Group (No Intervention): Control Group (CG) The CG received physiotherapy, exercises and education as per current standards of practice in our institution up until hospital discharge. Following discharge no further specific input or education was provided. Participants were contacted at least once during the study period to check on their general well being and to encourage attendance at the second assessment by the physiotherapy team. In line with the ethical requirements for the study, all control subjects were offered the chance to participate in the rehabilitation programme once their trial participation was completed following second assessment.

INTERVENTIONS:
Other: Rehabilitation Class — A 6 week programme of exercise and education in an out patient setting
  Arms: Treatment Group

SUMMARY:
Admission to an intensive care unit (ICU) due to illness has been shown to have a dramatic effect on the human body and mind. Following discharge from an ICU, patients suffer from varying degrees of weakness and muscle wasting. It can take many months before their strength returns to something like before they were ill. This weakness can have important consequences on an individual, affecting their ability to perform routine tasks (e.g. housework, shopping), and whether they can return to work or not. Not surprisingly, this inability to perform activities they used to do prior to their illness can have knock on effects on their mental well being and confidence.

What the investigators hope to see through this study is whether or not patients can recover their ability to perform exercise more quickly following an ICU admission if they undergo an exercise-based rehabilitation programme. The investigators also hope to see whether taking part in a rehabilitation programme has any affect on physical and mental well being.

The investigators hope to use a simple exercise test on a bicycle to assess subjects ability to exercise shortly after leaving hospital. We will then repeat the test after a period of physiotherapy lead rehabilitation to see if they have received any benefit from the programme. The investigators hope to show that by undergoing an exercise-based rehabilitation programme subjects will recover their ability to exercise more quickly than those who do not.

By means of questionnaires the investigators hope to see what effect the rehabilitation programme has had on participants physical and mental well being.

ELIGIBILITY:
Inclusion Criteria:

All patients over the age of 18

* admitted to a single, tertiary centre United Kingdom general intensive care unit (ICU)
* Invasively ventilated ≥ 5 days

Exclusion Criteria:

* Physical condition resulting in an inability to perform a cardio-pulmonary exercise test (CPET) or to participate in the rehabilitation classes,
* Psychiatric condition or impairment not allowing informed consent or compliance with the rehabilitation programme,
* Participation in an alternative rehabilitation programme,
* Terminal illness
* Poorly controlled cardio-respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Testing | At recruitment (within 6 weeks of hospital discharge) and then reassessed 8-10 weeks later
  Primary outcome was the change in exercise capacity measured by changes in peak VO2 and anaerobic threshold (AT) assessed using cardio-pulmonary exercise testing (CPET).

SECONDARY OUTCOMES:
Short Form 36 Health Questionnaire | At recruitment (within 6 weeks of hospital discharge) and then reassessed 8-10 weeks later
  Secondary outcome measures were changes in health related Quality of life (QoL). assessed using the Medical Outcome Study Short Form-36 questionnaire Version 2 (SF36v2). Subjects were asked to answer questions based on a 2-week recall period.